CLINICAL TRIAL: NCT02776969
Title: A Strategy to Search for Genes Predisposing to Papillary Carcinoma of the Thyroid When Mutated
Brief Title: A Gene Hunting Study for Familial Papillary Thyroid Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Matthew Ringel, Principal Investigator, Ohio State University Comprehensive Cancer Center
Other Study IDs: OSU-9812
Record Dates: First submitted 2016-05-12; First posted 2016-05-19 (Estimated); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Thyroid
Keywords: Papillary Carcinoma; Gene Hunting; Familial
MeSH Terms: conditions — Thyroid Diseases; Carcinoma, Papillary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, RNA, and (in some cases) lymphoblastoid cell lines will be maintained in the Ohio State University (OSU) Division of Human Genetics Sample Bank for the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this project is to identify genetic risk factors associated with familial papillary thyroid carcinoma (PTC). Papillary thyroid cancer is a type of cancer that shows high heritability. However, the specific genetic factors that cause an increased risk have been elusive.

DETAILED DESCRIPTION:
The aim of this project is to identify genetic risk factors associated with familial papillary thyroid carcinoma (PTC). This can be accomplished in several ways, including loss of heterozygosity studies as well as comparative gene expression analysis. When possible, linkage analysis on families with multiple individuals affected with PTC may also help identify the putative gene(s).

Study participants will be asked to:

1. Complete family history and medical history questionnaires
2. Sign a medical record release so that thyroid cancer pathology reports can be obtained
3. Supply a blood or saliva sample for genetic studies
4. Provide study related information to family members who are needed for family studies

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of PTC and a family history of PTC in 3 or more living relatives
* Affected and unaffected family members of the proband*

  * For familial cases (families with 4 or more cases of PTC), participation will be offered to all living family members with PTC or benign thyroid disease as well as selected unaffected first and second degree relatives. Participation may also be offered to spouses when needed for analyzing parent/offspring samples.

Exclusion Criteria:

* Known germline predisposition (ex: pathogenic PTEN variant)
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Families with at least 4 living individuals with a diagnosis of papillary thyroid carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 1998-08-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Genetic variants associated with familial papillary thyroid cancer as assessed by multiple genetic testing methodologies | Up to 5 years
  Variants will be assessed for segregation within families, expression in the normal thyroid and/or thyroid cancer, and functional significance

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Ringel, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu